CLINICAL TRIAL: NCT02264275
Title: The Influence of Aerobic Exercise Training on Disease Symptoms, Cardiovascular Fitness, Depression, Sleep and Quality of Life in Children and Adolescents Suffering From Inflammatory Bowel Disease in Switzerland
Brief Title: Influence of Aerobic Exercise Training (AET) on Inflammatory Bowel Disease (IBD) in Children and Adolescents
Acronym: Ex-CED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Basel (Other)
Collaborators: University Children's Hospital Basel (Other); Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Principal Investigator, Catherine Elliot, Dr. Catherine Elliot, University of Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DSBG-UniBasel-Ex-CED-2014-220
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Ulcerative Colitis; Crohn Disease; Depression; Sleep; Quality of Life; Motor Activity
Keywords: Aerobic Exercise; Exercise; Exergame; Behavior; Video Game; Inflammatory Bowel Disease; Children; Adolescents; Pediatric; Physical Fitness
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Depression; Motor Activity; Behavior; Inflammatory Bowel Diseases | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aerobic Exercise Training (Experimental): An 8-week Nintendo Wii at-home dancing exergame Intervention
  Interventions: Behavioral: Aerobic Exercise Training

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — The aerobic exercise training uses a television attached to a Nintendo Wii videogame console with a dance game to be played by participants on 5 days per week using a ramped-duration schedule (from 10-30 minutes of moderate physical activity daily).
  Other Names: Nintendo Wii; Exergame; Dance Videogame

SUMMARY:
The purpose of this study is to determine if aerobic exercise training can serve as comprehensive palliative care, whereby enhancing cardiovascular fitness, mitigating depressive symptoms and augmenting sleep while bolstering health related quality of life in youth with Crohn's Disease and Ulcerative Colitis.

DETAILED DESCRIPTION:
An AET intervention is designed to increase the aerobic fitness levels of IBD sufferers through daily activity, which is notably lower in this population and could be beneficial for sufferers managing this lifelong disease. With an increase in physical activity, the exergame aims to introduce, instill and integrate daily physical activity in the lives of IBD sufferers. The Just Dance Kids exergame for Nintendo Wii employs moderate intensity physical activity and is well suited for this study. The exergame intervention protocol will comprise a ramped duration aerobic exercise training starting with 10 minutes in week 1 and rises to 30 minutes per session in weeks 5 through 8. Just Dance Kids will be used by participants under the age of 11 and Just Dance for participants over the age of 10 due to the age appropriate dancing skill required in each game. The aim is to determine if this moderate intensity, 5 times per week exercise could decrease IBD flare-ups, improve cardiovascular fitness, reduce depressive symptoms, improve quality and quantity of sleep and improve the health-related quality of life in children and adolescents with IBD.

ELIGIBILITY:
Inclusion Criteria:

* aged 7 through 20 at start of study
* willing and able to volunteer in the study
* able to communicate and to complete questionnaires in German
* have a functioning television with Nintendo Wii compatibility at home
* provide participant written informed consent (when ≥11 years old at start of study)
* provide parental/legal caregiver written informed consent (when participant is ≤17 years old at start of study)
* provide oral informed consent (when ≤10 years old at start of study)

Exclusion Criteria:

* refusal to give necessary oral or written informed consent by patient and/or parent (legal caregiver)
* not aged 7 through 20 at start of study
* not willing and able to volunteer in the study
* has sibling enrolled in this study
* has severe physical diseases of the locomotor apparatus, psychotic disorders, severe affective disorders, eating disorders, mental retardation, autism spectrum disorder
* inability to communicate and complete questionnaires in German
* does not own a functional and Nintendo Wii-compatible television at home
* among female adolescents, pregnancy, breastfeeding or intention to get pregnant during the study
* has clinically significant cardiovascular disease
* enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Pediatric Disease Activity Index | 8 Weeks
  Uses either Crohn's Disease or Ulcerative Colitis Disease Activity Index respective to the patient's disease

SECONDARY OUTCOMES:
Sleep | 8 Weeks
  Uses Insomnia Severity Index and Daily Sleep Log
Depressive Symptomology | 8 Weeks
  Uses Child-S or Des-Teen with respect to participants age
Health Related Quality of Life | 8 Weeks
  KIDSCREEN-27
Estimation of Vo2Max | 8 Weeks
  Uses the Astrand-Rhyming cycle ergometer protocol

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Elliot, Dr. phil., Principal Investigator — University of Basel
Locations (3):
- Switzerland (3):
  - Universitäre Psychiatrische Kliniken Basel (UPK), Basel, Canton of Basel-City
  - Universitäts-Kinderspital beider Basel (UKBB), Basel, Canton of Basel-City
  - Universität Basel (Departement für Sport, Bewegung und Gesundheit), Basel, Canton of Basel-City

REFERENCES:
- [Derived] Mahlmann L, Gerber M, Furlano RI, Legeret C, Kalak N, Holsboer-Trachsler E, Brand S. Psychological wellbeing and physical activity in children and adolescents with inflammatory bowel disease compared to healthy controls. BMC Gastroenterol. 2017 Dec 12;17(1):160. doi: 10.1186/s12876-017-0721-7. PMID 29233119
- [Derived] Mahlmann L, Gerber M, Furlano RI, Legeret C, Kalak N, Holsboer-Trachsler E, Brand S. Impaired objective and subjective sleep in children and adolescents with inflammatory bowel disease compared to healthy controls. Sleep Med. 2017 Nov;39:25-31. doi: 10.1016/j.sleep.2017.08.015. Epub 2017 Sep 21. PMID 29157584
- See also: University of Basel, Department for Sport, Exercise and Health — https://dsbg.unibas.ch/
- See also: University of Basel Childrens Hospital — http://www.ukbb.ch/